CLINICAL TRIAL: NCT07003880
Title: Inhaled Methoxyflurane for In-Office Procedures in Otolaryngology
Brief Title: Penthrox in Otolaryngology
Acronym: PenthroxOTL
Status: Not yet recruiting | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-4462
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: All Adult Patients Undergoing an Otolaryngology Procedure With Inhaled Methoxyflurane as an Adjunct to Topical or Local Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing an otolaryngology in-office procedure using methoxyflurane: All adult patients undergoing any of the following procedures with inhaled methoxyflurane as an adjunct to topical or local anesthesia:
  * Skin lesion excision or reconstruction
  * Fine or core needle aspiration biopsy
  * Mucosal biopsy
  * Laryngeal injection or biopsy
  * Myringotomy with or without tympanostomy tube insertion
  * Inferior turbinate reduction
  * Septal button insertion
  Interventions: Drug: Methoxyflurane anesthesia

INTERVENTIONS:
Drug: Methoxyflurane anesthesia — A single Penthrox (3mL) self-inhaler will be administered 5-minutes prior to the onset of the procedure, before local anesthesia. Patients will undergo the procedure, have post-procedural vital signs, and remain in clinic for observation for 30 minutes post-procedure per our usual post-procedure monitoring.

SUMMARY:
Our objective is to explore the use of methoxyflurane anesthesia as an adjunct analgesic to local anesthesia during in-office otolaryngology procedures in a prospective pilot study. The main outcome of this study will be patient satisfaction with the medication and analgesia. Secondary outcomes will include level of sedation and analgesia, patient-reported post-procedural pain levels, and any reported adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing any of the following procedures with inhaled methoxyflurane as an adjunct to topical or local anesthesia:

  * Skin lesion excision or reconstruction
  * Fine or core needle aspiration biopsy
  * Mucosal biopsy
  * Laryngeal injection or biopsy
  * Myringotomy with or without tympanostomy tube insertion
  * Inferior turbinate reduction
  * Septal button insertion

Exclusion Criteria:

* Patient unable to complete the post-procedure questionnaire (either due to time constraints, neurocognitive impairment, etc.)
* Presence of any contraindications to inhaled methoxyfluorane per product monograph:

  * Patients less than 18 years of age
  * Pregnancy, intended pregnancy, or current breast-feeding
  * Inadequate patient understanding or lack of cooperation
  * Decreased level of consciousness or head injury
  * History of clinically significant renal impairment, e.g., reduced renal output
  * History of liver dysfunction following previous exposure to halogenated anesthetics
  * Current use of tetracycline antibiotics
  * Personal or genetic history of malignant hyperthermia
  * Muscular dystrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing an otolaryngology proceure in the Otolaryngology clinic of the Jewish General Hospital with inhaled methoxyflurane as an adjunct to topical or local anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
TSQM-1.4 (Treatment Satisfaction Questionnaire for Medication 1.5) | At first follow-up visit (within 1 month post-procedure)
  This is a validated 14-item including Likert scales and dichotomous (yes/no) items on the effectiveness, side effects, convenience and global satisfaction with the medication taken

SECONDARY OUTCOMES:
Ability to complete intended procedure | At procedure visit
  Documented by clinic nurse post- procedure
Modified Ramsay Sedation score | At procedure visit
  Maximal sedation score during procedure documented by clinic nurse
Adverse events | At procedure visit and first follow-up visit (within 1 month post-procedure)
  Either self- or physician-reported
Visual analog pain scale | At procedure visit
  Maximal degree of pain during procedure